CLINICAL TRIAL: NCT02119000
Title: Comparison of Two Types of Bowel Preparation for Inpatient Colonoscopy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty in recruitment
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Alan Barkun, Gastroenterologist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: GEN 13-148; GEN 13-148
Record Dates: First submitted 2014-01-26; First posted 2014-04-21 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Hospitalized Patients
MeSH Terms: interventions — Bisacodyl

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEG electrolytes 2L/2L split dose (Experimental)
  Interventions: Drug: PEG/electrolytes 2L/2L split dose
- Bisacodyl 15 mg and PEG/electrolytes 1L/1L split dose (Active Comparator)
  Interventions: Drug: Bisacodyl 15 mg and PEG/electrolytes 1L/1L split dose

INTERVENTIONS:
Drug: PEG/electrolytes 2L/2L split dose — Polyethylene glycol 17gm X 4 At 18h00 the day prior the colonoscopy, dilute 2 sachets in 2 L of water and drink 240 mL every 10 minutes On the day of the procedure, 4-5 hours prior the colonoscopy, dilute 2 sachets in 2 L of water and drink 240 mL every 10 minutes
  Arms: PEG electrolytes 2L/2L split dose
Drug: Bisacodyl 15 mg and PEG/electrolytes 1L/1L split dose — Bisacodyl 15 mg x 3
  At 14h00 the day prior the endoscopic procedure: take 3 tablets of Bisacodyl ER (15 mg) orally then 5 hr later:
  PEG/electrolytes 1L/1L Polyethylene glycol 17gm Dilute one sachet of Polyethylene glycol 17gm in 1 L of water Start drinking at around 19h00 the night prior the colonoscopy Drink 240 ml every 10 minutes The day of the colonoscopy. At (4 hrs prior the procedure). Dilute on sachet of PEG and drink 240 ml every 10 minutes
  Arms: Bisacodyl 15 mg and PEG/electrolytes 1L/1L split dose

SUMMARY:
Bowel preparation is a crucial step prior to colonoscopy to help with the optimal assessment of the colonic mucosa. Inadequate bowel preparation increases the length of the procedure, and is associated with decreased lesional detection rates. The ideal bowel preparation formulation should be able to completely clean the bowel, without leaving solid or liquid residues, and without modifying the mucosal appearance.

Bowel preparation may be administered in hospitalised patients or in the ER. Patients have less control on their environment and the intake of the bowel preparation. For example, there may be a delay in pharmacy delivery or inadequate supervision by the treating personnel. Hospitalised patients have more comorbidities, are usually less autonomous and mobile - both can add to the barriers leading to an adequate bowel preparation. Multiple studies have identified hospitalization status as an independent risk factor for poor bowel preparation.

The objective of this study is to access which bowel preparation regimen, between PEG 3350 with electrolytes 2L the day before and 2L the day of the colonoscopy vs bisacodyl + PEG 3350 with electrolytes 1L the day before and 1L the day of the colonoscopy, results in the cleanest bowel preparation in hospitalised patients.

ELIGIBILITY:
Inclusion Criteria

* 18 years or older
* Be able to comprehend the trial and provide written informed consent in French or English, or a close relative with power of attorney
* Have a recognised indication for full colonoscopy after evaluation by a gastroenterologist or surgeon
* Be hospitalized or in the ED of a participating hospital center.
* Need to receive a bowel preparation during hospitalization or the ED stay.
* Be able to complete the follow-up patient response form in French or English

Exclusion Criteria:

* Patient refusal
* A suspected or diagnosed bowel obstruction
* A toxic megacolon
* Ileus
* Decompensated heart failure
* Severe acute renal failure
* Severe electrolyte imbalance
* Previous bowel preparation in the last 7 days
* Pregnancy
* Time of randomization before 9h00 or after 22h00

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2015-08; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Efficacy | following colonoscopy
  Which bowel preparation regimen, between PEG 3350 with electrolytes 2L the day before and 2L the day of the colonoscopy vs bisacodyl + PEG 3350 with electrolytes 1L the day before and 1L the day of the colonoscopy, results in the cleanest bowel preparation in hospitalised patients.

SECONDARY OUTCOMES:
Tolerability | Before colonoscopy
  A questionnaire will be used to assess which is the most tolerable and acceptable to patients between the two bowel preparation regimens
Clinical quality standards | After colonoscopy
  Does the bowel preparation given prior to in-hospital colonoscopy result in an excellent or good preparation rate that falls within the required clinical quality standards?
Cecal/ileal intubation rate | Following colonoscopy
  What is the cecal/ileal intubation rate for colonoscopies performed in hospitalized patients?
Polyp detection rate | Following colonosopy
  What is the polyp detection rate for colonoscopies performed in hospitalized patients?

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - McGill University Health Centre, Montreal, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec